CLINICAL TRIAL: NCT05925868
Title: The Mental Health Effects of a Mindfulness App in Parents of a Child With Medical Complexity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boise State University (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Cara Gallegos, Associate Professor, Boise State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 186-SB22-056
Record Dates: First submitted 2022-09-28; First posted 2023-06-29 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Depression; Family Dynamics; Stress, Psychological; Chronic Illness; Parents
Keywords: mindfulness app; parents; child with chronic illness; stress; depression; family management; Headspace
MeSH Terms: conditions — Depression; Stress, Psychological; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile app (Experimental): Parents will be given access the Headspace, a mobile mindfulness app, and instructed to use it at least 4 days a week for a minimum of 10 minutes
  Interventions: Behavioral: mindfulness app

INTERVENTIONS:
Behavioral: mindfulness app — Parents will use the mindfulness app, Headspace, for at least 10 minutes on 4 days/week.
  Other Names: Headspace

SUMMARY:
The number of children with special health care needs (CSHCN) in the US is nearly 20% of children representing approximately 14.6 million children nationally. A subgroup of CSHCN are children who have the most intensive healthcare needs known as children with a medical complexity (CMC). Parents of CMC experience many challenges. In addition to typical caregiver tasks, parents of a CMC may experience added stress and are more likely to experience higher rates of anxiety, depression, and post-traumatic stress disorder than parents of healthy children. This project aims to explore the acceptability and feasibility of a mindfulness mobile application for parents of a CMC as well as determine the effectiveness of mindfulness application use on stress, depression, and family management in parents of a CMC. Forty-five participants will be recruited and given access to a mindfulness application and instructed to use it at least 4 days a week for at least 10 minutes. Parents will fill out questionnaires on app usage, as well as stress, depression, and family management. This work will be accomplished through a pilot single arm approach.

DETAILED DESCRIPTION:
Significance The prevalence of pediatric chronic conditions is increasing rapidly. Medical advances in the last half-century created a dramatic change in the prevalence of childhood-onset diseases leading to a growing number of CSHCN, increasing >400% since the 1960s.The estimated prevalence of CMC ranges from 1% to 5% or approximately 680,000 children depending on the definition. The majority of parents function as unlicensed caregivers in managing life-sustaining technologies and administering medications and caring for their CMC as well as their other well children in the household. Parents of CMC experience worse mental and physical health outcomes compared to parents of healthy children. They face many challenges such as difficulty accessing medical and nonmedical services and financial problems related to costs associated with the child's care. It is well documented that these parents experience high levels of stress and depression. 60% of parents of a child with chronic illness experience depression compared to 10% in mothers of healthy newborns. Parents of CMC are at higher risk for experiencing suboptimal mental health outcomes over time. In addition to poor psychological outcomes, parent caregivers also experience worse physical health such as low back pain due to lifting, migraine headaches, chronic fatigue, sleep deprivation, and stomach/intestinal ulcers. Although not specifically studied in parents of CMC, a recent systematic review found that the effects of stress included poor general physical health, increased pain and disability, lower quality of life, and higher risk of all-cause mortality.

While psychological interventions have been shown to improve parent distress, parenting behaviors, and family conflict in parents of a CSHCN, less is known about parents of a CMC. These parents often have significant and diverse needs and benefit from specific, targeted interventions. Previously tested interventions include: parenting programs, targeted parent behavior change such as cognitive behavioral therapy, peer support, psychological interventions, resourcefulness training. Other studies indicate that improving psychological outcomes of caregivers affects emergency room visits and hospitalizations. Parents of CMC often lack the resources to obtain assistance. This will be one of the first studies to examine a simple, cost-effective intervention that parents can access from their home. Future studies aimed at understanding the physical and psychological effects and benefits of a mindfulness app are important for this vulnerable population.

Innovation The research is novel in its approach of examining the feasibility and acceptability of a mindfulness app in parent caregivers of this vulnerable population of CMC for a period of 28 days. Mindfulness meditation delivered in a traditional format (i.e., 8 weekly in-person 60-90 minute sessions) has become a popular practice to improve mental health with several researchers reporting a decrease in depressive symptoms, stress, and anxiety in parents of a child with chronic illness. Despite these benefits, traditional mindfulness programs can be difficult to access because they are time and cost-intensive. Mobile applications (apps) for smartphones present an opportunity to overcome barriers associated with typical mindfulness meditation programs. There are several popular mindfulness apps available. One of the most widely used apps, Headspace®, offers hundreds of hours of instructor-guided meditation exercises. Mindfulness app use has benefited users in as little as 10 days but is often studied for 28 days. Although there is significant research demonstrating the effectiveness of mindfulness programs delivered through a mobile app in other populations, to the investigator's knowledge, there is no research examining the use and efficacy in parents of CMC.

Approach Research Design. The proposed study is a single arm pilot study to explore the feasibility, acceptability and efficacy of the intervention and to identify intervention and protocol challenges prior to development of a RCT.

Inclusion/Exclusion criteria. Inclusion criteria are parents: 1. 18 years or older of a child with medical complexity, 2. with daily access to a mobile device (i.e. smartphone or tablet), 3. score > 4 on Perceived Stress Scale-4 (PSS-4), and 4. able to read English (the mindfulness app is only available in English). Exclusion criteria: a current mindfulness practice (i. e., practice ≥15 min per day of meditation or yoga within the past 6 months).

Recruitment. Forty-five participants will be recruited from a local non-profit organization and local community hospital's pediatric specialty outpatient clinic. The non profit supports approximately 115 families and the pediatric clinics oversee the care of approximately 4,000 CMC throughout the state of Idaho. An informational flyer will be distributed to families in the pediatric specialty clinic patient waiting areas. The flyer will have a link and QR code to the enrollment forms including a questionnaire to screen for eligibility and a copy of the consent form with the study procedures. The two sites will provide an opportunity for increased recruitment and sample diversity. For this pilot study, 45 participants will allow for potential attrition and a sufficient number to meet the pilot study aims and provide an effect size for a power analysis in larger studies. The investigators believe that the study team can successfully manage 45 participants with initial contact, weekly and end-of-study follow-up.

Consent. Participants will email the consent forms to the PI after reading the study procedures.

Intervention. Once the consent form is returned, the PI will assign a number to the participant. This spreadsheet will have their name, email address, and cellphone number. It will be stored electronically and separate from the consent forms in a secure, password protected. The PI will send the participants an electronic link to fill out the baseline study questionnaires. Upon completion, the research assistant will send the participants a code and directions to download the mindfulness app, Headspace®. Headspace was selected because it had the highest average rating (4.0 out of 5) in a review of 23 mindfulness apps. A confirmatory text message will be sent to participants reminding them which program to start and to use the app at minimum 4 days per week for at least 10 minutes for four weeks. Participants will be asked to work through the Basic course 1, 2, and 3 consisting of 10 sessions ranging from 4 minutes to 11 minutes, each. The basic course provides the fundamentals of meditation and mindfulness. In the Basics 2 course, participants start to deepen their practice, and in the Basic 3 course, they will apply mindfulness to everyday life. If participants complete the Basic courses, they will be asked to continue using the app, but can choose optional classes from the Headspace library. The undergraduate research assistant will send weekly text message reminders to encourage participant app use.

Data collection. Each week, the undergraduate research assistant will send out the appropriate questionnaires to participants. All data will be collected using Qualtrics via an email link. Participants will be able to complete the surveys at a time that is convenient and a location that is comfortable for them. Participants will receive a $75 Amazon gift card for completing the baseline and the Week 4 questionnaires. Instruments. For Aim 1, participants will complete a brief weekly engagement and enjoyment questionnaire by providing the total number of Headspace app minutes and programs used. At the end of the 4 week intervention, parents will complete a questionnaire on feasibility and acceptability. For Aim 2, participants will complete stress, depression, and family management surveys at baseline and at the end of the 4 week intervention (approximately 25 minutes to complete all instruments at baseline and week 4). In addition, participants will complete brief, weekly stress and engagement/enjoyment instruments that should take less than 5 minutes to finish (Table 1). The following questionnaires will be used:

Demographics. Participants will complete a demographic questionnaire to examine parent demographics (i.e., age, gender, income, education, occupation) and child clinical variables (i.e., age, number of providers seen, diagnosis, time since diagnosis).

Stress. The Pediatric Inventory for Parents (PIP) is a 42-item self-report tool that was developed to measure parenting stress related to caring for a child with a chronic illness.

Depression. The Patient Health Questionnaire (PHQ-9) is a 9-item self report tool that was developed to measure the severity of depression. For each question, participants rate their level of feeling on a scale of 0 - 3 (0 = not at all; 3 = nearly every day).

Family Management. The Family Management Measurement (FaMM) is a 45-item questionnaire used to measure how parents manage the care of their child with a chronic illness.

Weekly Stress Questionnaire. The Perceived Stress Scale (PSS-10), a 10-item questionnaire used to assess stress, has been used in a variety of populations. The total scale scores range from 0 to 40; higher scores indicate more perceived stress.

Usage and Enjoyment Questionnaire. This is based on a previous questionnaire and consists of closed-ended questions such as, how many minutes they used the app, what programs they used, and to what extent the activities were enjoyable or difficult to complete.

Feasibility and Acceptability Questionnaire. This is based on a previous questionnaire. It consists of closed-ended and open-ended questions that ask parents to rate the app, whether they would recommend it, and asks about their experience using the app and whether they intend to continue its use.

Data management and analysis. The surveys will be administered online via Qualtrics. Confidentiality will be maintained by storing all data on a password protected server maintained by Boise State University. Only study personnel will have access to the data. The investigators will address analysis of Aim 1 with descriptive statistics from the Feasibility and Acceptability and the Usage and Enjoyment questionnaires. Investigators will employ content analysis of responses to the open-ended questions from the Feasibility and Acceptability questionnaire to develop themes. For analysis of Aim 2, descriptive statistics will be used to describe parent stress, depression and family management. To address the hypotheses in Aim 2, the investigators will use repeated measures ANOVA in a mixed model framework to identify changes in stress, depression, and family management indices, controlling for weekly usage minutes. Additional covariates of weekly stress, app enjoyment, and baseline demographics may also be examined as covariates in this model. The need for propensity score weighting will be evaluated. The assessment of study dropouts, and the extent to which these participants may bias the overall statistical findings, will be conducted at the outset of the data analysis. In addition to ensuring model validity, these analyses will help identify barriers for this population in using the app or participating in mindfulness-based stress reduction in general.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older of a child with medical complexity with daily access to a mobile device (i.e. smartphone or tablet)
* score > 4 on Perceived Stress Scale-4 (PSS-4)
* able to read English (the mindfulness app is only available in English).

Exclusion Criteria:

- a current mindfulness practice (i. e., practice ≥15 min per day of meditation or yoga within the past 6 months).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of a mindfulness mobile application for parents of a CMC | 4 weeks
  The feasibility scale will be used to assess the feasibility of the app during and after the study. This is based on a questionnaire by Rung, Oral, Berghammer, Peters (2020)35. It consists of closed-ended and open-ended questions that ask parents to rate the app, whether they would recommend it, and asks about their experience using the app and whether they intend to continue its use.
To describe the efficacy of a mindfulness app on stress in parents of a child with CMC | 4 weeks
  The Pediatric Inventory for Parents (PIP) will be used to assess stress before and after mindfulness app use. The PIP has 42 questions, scored 1-5 with higher scores indicating higher stress.
To describe the efficacy of a mindfulness app on depression | 4 weeks
  The PHQ-9 will be used to describe the effects of a mindfulness app on depression scores. The PHQ includes 9 questions ranging from 0-3 with higher numbers indicating a higher depression score.
To describe the efficacy of a mindfulness app on family management | 4 weeks
  The Family Management Measure (FaMM) will be used to describe the effects of a mindfulness app on family management. There are 45 items, ranging from 1-5 with higher scores indicating higher difficulty with family management

CONTACTS AND LOCATIONS:
Overall Officials: Cara Gallegos, PhD, BSN, Principal Investigator — Boise State University
Locations (1):
- St. Luke's Regional Hospital, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD and the study protocol will be made available to investigators who contact the PI.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available after data has been collected.
Access Criteria: Requests will be reviewed by the PI. IRB and a data transfer agreement will be required

DOCUMENTS (1):
  • Informed Consent Form (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT05925868/ICF_000.pdf